CLINICAL TRIAL: NCT00752258
Title: A Phase III, Multi-Center, Long-Term, Repeat-Treatment, Open-Label, Single-Arm Trial to Demonstrate the Safety of Repeat Treatment With PurTox® for the Treatment of Glabellar Rhytides ("Frown Lines")
Brief Title: A Long-Term Safety Study of Repeat Treatment With PurTox® for Frown Lines Between the Eyebrows
Acronym: PT-03c
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mentor Worldwide, LLC (Industry)
Collaborators: Synteract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-03c
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Glabellar Rhytides
Keywords: Botulinum Toxin Type A; Botulinum Toxin; Glabellar Rhytides; Rhytides; Frown Lines; Neuromuscular Agents; Neurotoxin; Forehead; Eyebrow; Wrinkle; Frown Lines Between the Eyebrows
MeSH Terms: interventions — Botulinum Toxins, Type A; Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Mentor Purified Toxin Botulinum Toxin Type A
  Interventions: Drug: Mentor Purified Toxin Botulinum Toxin Type A

INTERVENTIONS:
Drug: Mentor Purified Toxin Botulinum Toxin Type A — All subjects will receive five 0.1 mL intramuscular injections (two in each corrugator and one in the procerus muscle) at each Treatment Visit. The total treatment dose (sum of the five injections) to be administered will be 30 U of Mentor Purified Toxin. Subjects will have many Treatment Visits throughout the course of the three-year study.
  Other Names: Botulinum Toxin Type A; Botulinum Toxin

SUMMARY:
The overall purpose of this study is to evaluate the long-term safety of repeat treatment with an intramuscular dose of Mentor Purified Toxin for the reduction of frown lines.

DETAILED DESCRIPTION:
This is a Phase III, multi-center, open-label study to evaluate the long-term safety of repeat treatment with PurTox for the treatment of glabellar rhytides. Up to 576 patients will be enrolled at 12 sites in the U.S.A. and some of these patients may have participated in Mentor Purified Toxin Phase I, II and IIIa studies. Safety and tolerability of the repeat treatment with Mentor Purified Toxin will be examined during the study.

Effectiveness will be determined by the degree of frown line reduction, during maximum forced frown and at rest (neutral expression):

* as assessed live by the study doctor,
* as assessed live by the subject, and;
* as assessed by an independent reviewer based on subject photographs

Frown lines are graded on level of severity based on this scale:

Severity

* Minimal (0)
* Mild (1)
* Moderate (2)
* Severe (3)

All subjects meeting the study eligibility criteria will be treated with 30 U of Mentor Purified Toxin. Following the treatment, follow-up assessments are scheduled as follows: telephone safety assessments on post-treatment Days 7 and 14, a clinic visit on post-treatment Day 30, and a telephone safety assessment on post-treatment Day 60 and monthly thereafter until re-treatment.

A subject will be re-treated when he/she attains grade 2 (Moderate) or 3 (Severe) in the investigator's and subject's ratings of the severity of glabellar rhytides at maximum frown on a 4-point categorical scale, but not earlier than 90 days following the prior treatment. The subject will call the site when he/she rates the glabellar rhytides as grade 2 or 3 in severity to schedule an appointment for re-evaluation and possible re-treatment. The appointment must occur within 2 weeks of the subject's call but not earlier than 90 days post the previous injection. If at the clinic visit the subject's glabellar rhytides are graded by the investigator as grade 2 or 3 in severity and other eligibility criteria are met (e.g., negative urine pregnancy test in female subjects of childbearing potential), the subject will be re-treated. If a subject is eligible for re-treatment on or before 90 days post the previous injection, he/she will receive treatment of Mentor Purified Toxin on or after 90 days. If a subject is not eligible for re-treatment at 90 days, he/she can return to the clinic monthly until attaining grade 2 (Moderate) or 3 (Severe) in the investigator's and subject's ratings of the severity of glabellar rhytides at maximum frown on a 4-point categorical scale, at which time he/she will receive another treatment of Mentor Purified Toxin.

If a subject chooses not to be re-treated with Mentor Purified Toxin when he/she becomes eligible for re-treatment, the subject will be followed up with the monthly telephone safety assessments and annual safety visits to the clinic. It is anticipated that most subjects will receive multiple repeat treatments during this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who are 18 years of age or older with an interest in the effacement of glabellar rhytides, with or without previous Botulinum Toxin Type A exposure;
2. In good physical and mental health as determined by the investigator based on medical history, physical examination, and/or clinical laboratory tests;
3. Noticeable presence of the glabellar rhytides for a period of 6 months or longer;
4. Score at least a 2 (moderate severity) at baseline screening on the investigator's and subject's assessments (reference photographs provided) at forced frown; and
5. Capable of understanding and complying with the protocol and must have signed the informed consent document prior to performance of any study-related procedures.

Exclusion Criteria:

1. A history of psychiatric problems that, in the investigator's opinion, is severe enough potentially to interfere with subject outcomes;
2. A history of autoimmune disease, that, in the opinion of the investigator, might interfere with subject outcomes (e.g., osteoarthritis is not considered an exclusion criterion; however, subjects with dermatomyositis are not permitted to participate in this study);
3. A history or presence of clinically significant cardiovascular, respiratory, hepatic/biliary, renal, gastrointestinal, endocrine, or neurological disorders constituting a possible risk factor that, in the investigator's opinion, is severe enough potentially to interfere with subject outcomes;
4. Inability to substantially efface glabellar lines by manually spreading skin apart;
5. Eyelid ptosis;
6. Myasthenia gravis or diseases of neurotransmission (from medical history);
7. Current history of facial nerve paralysis;
8. Concurrent dermatologic disease of the face in the glabellar area that is deemed by the investigator to make the subject an inappropriate candidate for the study;
9. Recent flu-like syndrome that, in the investigator's opinion, is severe enough potentially to interfere with subject outcomes;
10. Neuromuscular disorder that, in the investigator's opinion, is severe enough potentially to interfere with subject outcomes;
11. Active multisystems disease that, in the investigator's opinion, might influence the outcome measures or the safety of the subject;
12. Has any condition(s) that in the investigator's opinion would a) warrant exclusion from the study, or b) prevent the subject from completing the study;
13. Currently receiving aminoglycoside antibiotic therapy, curare-like drugs, quinidine, succinylcholine, polymyxins, anticholinesterases, magnesium sulfate, or lincosamides;
14. Has taken any investigational drug during the 30 days prior to screening visit;
15. Have had dermal filler treatment to glabellar area during the 6 months prior to screening visit;
16. Female subjects who are pregnant or lactating. Female subjects who are of childbearing potential must have negative urine pregnancy test results prior to enrollment into the study. Such subjects, including peri-menopausal women who have had a menstrual period within one year, must be using appropriate birth control (see protocol/informed consent for description);
17. Unwilling or unable to comply with the protocol or to cooperate fully with the investigator and site personnel; or
18. Unable to understand verbal and/or written English or any other language in which a certified translation of the informed consent document is available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Estimation of the incidences of treatment-emergent adverse events, serious treatment-emergent adverse events, and treatment-emergent laboratory abnormalities, when PurTox is administered in repeated treatments. | Throughout

SECONDARY OUTCOMES:
Estimate across treatment cycles the frequency with which subjects are responders at Day 30, based on an assessment of rhytide severity at maximum frown of 0 or 1 by the investigator | Day 30/Across all Treatment Cycles
Estimate across treatment cycles the frequency with which subjects are responders at Day 30, based on an assessment of rhytide severity at maximum frown of 0 or 1 by the subject | Day 30/Across treatment all cycles
Estimate across treatment cycles the frequency with which subjects are responders at Day 30, based on assessments of rhytide severity at maximum frown of 0 or 1 by both the investigator and the subject | Day 30/Across all treatment cycles
Estimate across treatment cycles the frequency with which subjects, who are responders at Day 30, based on subject assessment at maximum frown, continue to be responders at Days 90, 120, 150, and 180. | Day 30 through Day 180/Across all treatment cycles

CONTACTS AND LOCATIONS:
Overall Officials: Corey Maas, Study Director
Locations (1):
- Mentor Worldwide, LLC, Santa Barbara, California, United States